CLINICAL TRIAL: NCT04411004
Title: Persistence of Rectal Endometriosis After Laparoscopic Shaving of Rectovaginal Endometriosis Infiltrating the Rectum
Brief Title: Persistence Disease After Laparoscopic Shaving of Rectal Endometriosis
Acronym: ENDO-SHAVING
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: ENDO-SHAVING
Record Dates: First submitted 2020-05-19; First posted 2020-06-01 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Endometriosis, Rectum
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who underwent shaving for rectal endometriosis
  Interventions: Diagnostic Test: Transvaginal ultrasound; Behavioral: 5-point Likert scale

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Transvaginal ultrasonographic scan to diagnosis the recurrence of rectal endometriosis
Behavioral: 5-point Likert scale — Subjective scale to evaluate satisfaction to previous surgical treatment for rectal endometriosis

SUMMARY:
When performing shaving of a rectal endometriotic nodule, the surgeon can use the macroscopic appearance of the nodule and the tactile feedback provided by the laparoscopic instruments to decide the area of the bowel that needs to be excised. Theoretically, compared with segmental bowel resection, the shaving technique may expose the patients to a higher risk of persistence of intestinal endometriosis. The objective of this ultrasonographic study was to assess the risk of rectal endometriosis persistence following laparoscopic shaving of rectovaginal nodules.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent laparoscopic shaving of rectovaginal endometriosis infiltrating the rectum

Exclusion Criteria:

* patients underwent previous bowel surgery (except appendectomy);
* patients experienced postoperative complications (such as pelvic abscess, rectovaginal fistula, ureteral injuries)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent shaving of rectal endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with rectal recurrence of endometriosis | 3 months after the surgical approach
  Evaluated by ultrasound
Number of patients with rectal recurrence of endometriosis | 6 months after the surgical approach
  Evaluated by ultrasound

SECONDARY OUTCOMES:
Satisfaction of patients to the previous surgical treatment | 3 months after the surgical approach
  Evaluated by five-point Likert scale
Volume of nodules in patients with rectal recurrence of endometriosis | 3 months after the surgical approach
  Evaluated by ultrasound
Satisfaction of patients to the previous surgical treatment | 6 months after the surgical approach
  Evaluated by five-point Likert scale
Volume of nodules in patients with rectal recurrence of endometriosis | 6 months after the surgical approach
  Evaluated by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alhayo S, Leonardi M, Lu C, Gosal P, Reid S, Barto W, Condous G. Ultrasound evaluation of pouch of Douglas obliteration and rectal deep endometriosis in women who have had previous combined colorectal and gynaecological laparoscopic surgery for rectal endometriosis: A pilot study. Aust N Z J Obstet Gynaecol. 2020 Apr;60(2):258-263. doi: 10.1111/ajo.13112. Epub 2020 Jan 9. PMID 31919838